CLINICAL TRIAL: NCT02375932
Title: Pre-Visit Prioritization for Complex Primary Care Patients With Diabetes
Brief Title: Pre-Visit Prioritization for Complex Patients With Diabetes
Acronym: PVP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CN-13-1579; R01DK099108 (NIH)
Record Dates: First submitted 2015-02-24; First posted 2015-03-03 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Electronic Medical Records; Primary Health Care; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-Visit Tool (Experimental): Patients whose primary care physicians are allocated to the intervention arm will receive a secure electronic message shortly after scheduling an appointment with their provider asking them to complete a pre-visit prioritization survey using the kp.org patient portal
  Interventions: Behavioral: Pre-Visit Tool
- Usual Care Control (Active Comparator): Patients whose primary care physicians are allocated to the control arm will continue with usual care
  Interventions: Behavioral: Usual Care Control

INTERVENTIONS:
Behavioral: Pre-Visit Tool — Patients receive a secure electronic message from their primary providers asking them to prepare for their visit by reviewing important areas of care and identifying their top priorities for discussion at a scheduled visit
  Arms: Pre-Visit Tool
Behavioral: Usual Care Control — Patients continue to receive usual care from their primary care provider
  Arms: Usual Care Control

SUMMARY:
Patients with type 2 diabetes are increasingly complex. Lack of time to address all patient and provider priorities during primary care visits represents a barrier to effective primary care. The investigators propose to design, implement, and evaluate in a randomized clinical trial a web-based tool linked to the electronic health record (EHR) that will enable complex patients to easily define care priorities for their upcoming visit.

DETAILED DESCRIPTION:
Patients with type 2 diabetes are increasingly living with multiple concurrent conditions and complicated medical regimens. For these patients, diabetes management decisions and treatment goals must be addressed within the larger context of other competing health concerns. In parallel, clinical advances have led to a substantial increase in the number of tasks that primary care providers must perform during each visit. These twin trends present a formidable challenge to effective diabetes primary care. We hypothesize that among complex patients not meeting diabetes management goals, a web-based health IT tool to help patients explicitly prioritize all health issues (both related and unrelated to diabetes) and then submit these priorities directly into the electronic health record (EHR) for a scheduled visit with their primary care provider will result in more effective diabetes management over time. To test this hypothesis, we propose to design, implement, and evaluate in a randomized clinical trial a web-based tool linked to the EHR that will enable complex patients to easily define care priorities for their upcoming visit.

ELIGIBILITY:
Primary care physicians (PCPs) at Kaiser Permanente Northern California with potentially eligible patients (type 2 diabetes and HbA1c > 8.0%) wil be recruited and consented to participate in this study. PCPs will review lists of potentially eligible patients of theirs (defined below). Patients approved by PCP's allocated to the intervention arm will be sent a secure message on the PCPs behalf asking them to review the Pre-Visit Prioritization Questionnaire to identify top priorities for discussion at the next scheduled visit.

Patient Inclusion Criteria:

* Current adult member (> 21 years old)
* Diagnosis of type 2 diabetes with most recent HbA1c > 8.0%
* English as primary language
* Registered on kp.org.

Patient Exclusion Criteria:

* Excluded by PCP, and/or: terminal illness, in hospice care or reside in a long-term care facility, severe mental illness (e.g. schizophrenia or personality disorder), currently or recently pregnant, and/or significant dementia

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2015-03; Primary Completion 2016-10-21 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Glycemic Control (HbA1c control (% patients < 7.0% and mean HbA1c levels) | 1 year after enrollment
  We will compare HbA1c control (% patients < 7.0% and mean HbA1c levels) between intervention and control arms

SECONDARY OUTCOMES:
Patient assessment of visit communication (measures of communication quality using validated instruments) | Shortly after visit with PCP
  We will call a subset of patients in the intervention and control arms after attending a visit with their PCP to assess measures of communication quality using validated instruments

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Grant, MD MPH, Principal Investigator — Division of Research, Kaiser Permanente Northern California

REFERENCES:
- [Background] Grant RW, Adams AS, Bayliss EA, Heisler M. Establishing visit priorities for complex patients: A summary of the literature and conceptual model to guide innovative interventions. Healthc (Amst). 2013 Dec;1(3-4):117-122. doi: 10.1016/j.hjdsi.2013.07.008. PMID 24944911
- [Result] Grant RW, Uratsu CS, Estacio KR, Altschuler A, Kim E, Fireman B, Adams AS, Schmittdiel JA, Heisler M. Pre-Visit Prioritization for complex patients with diabetes: Randomized trial design and implementation within an integrated health care system. Contemp Clin Trials. 2016 Mar;47:196-201. doi: 10.1016/j.cct.2016.01.012. Epub 2016 Jan 26. PMID 26820612
- [Result] Zamudio CD, Sanchez G, Altschuler A, Grant RW. Influence of Language and Culture in the Primary Care of Spanish-Speaking Latino Adults with Poorly Controlled Diabetes: A Qualitative Study. Ethn Dis. 2017 Dec 7;27(4):379-386. doi: 10.18865/ed.27.4.379. eCollection 2017 Fall. PMID 29225438
- [Result] Grant RW, Altschuler A, Uratsu CS, Sanchez G, Schmittdiel JA, Adams AS, Heisler M. Primary care visit preparation and communication for patients with poorly controlled diabetes: A qualitative study of patients and physicians. Prim Care Diabetes. 2017 Apr;11(2):148-153. doi: 10.1016/j.pcd.2016.11.003. Epub 2016 Dec 1. PMID 27916628
- [Derived] Vo MT, Uratsu CS, Estacio KR, Altschuler A, Kim E, Alexeeff SE, Adams AS, Schmittdiel JA, Heisler M, Grant RW. Prompting Patients with Poorly Controlled Diabetes to Identify Visit Priorities Before Primary Care Visits: a Pragmatic Cluster Randomized Trial. J Gen Intern Med. 2019 Jun;34(6):831-838. doi: 10.1007/s11606-018-4756-4. Epub 2019 Feb 11. PMID 30746642